CLINICAL TRIAL: NCT02893553
Title: The Effects of Normalizing Blood Pressure on Cerebral Blood Flow in Hypotensive Individuals With Spinal Cord Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Jill M. Wecht, Ed.D., Research Health Scientist, James J. Peters Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WEC-16-015
Record Dates: First submitted 2016-08-29; First posted 2016-09-08 (Estimated); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Spinal Cord Injury; Autonomic Dysreflexia; Baroreceptor Integrity; Sympathetic Integrity; Vagal Integrity; Autonomic Integrity; Hypotensive; Cognitive Function; Cerebral Blood Flow; Blood Pressure
MeSH Terms: conditions — Spinal Cord Injuries; Autonomic Dysreflexia | interventions — Midodrine; Pyridostigmine Bromide; mirabegron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study 1 (Experimental): Study 1: is a dose escalation to determine the individualized dose of each of 3 medications (midodrine, pyridostigmine, mirabegron) that increases SBP into the normal range (111-139 mmHg). The investigator will be using midodrine hydrochloride, pyridostigmine bromide and mirabegron.
  Interventions: Drug: Midodrine Hydrochloride; Drug: Pyridostigmine Bromide; Drug: Mirabegron
- Study 2 (Experimental): Study2: is a randomized placebo-controlled double-blinded investigation to determine the effect of the normalization of SBP on cerebral blood flow, cognitive function (memory and attention processing) and quality of life. The investigator will be using midodrine hydrochloride, pyridostigmine bromide, mirabegron and placebo.
  Interventions: Drug: Midodrine Hydrochloride; Drug: Pyridostigmine Bromide; Drug: Mirabegron; Other: Placebo

INTERVENTIONS:
Drug: Midodrine Hydrochloride — study 1 will be single blind. study 2 will be blinded randomized-control trial.
  Other Names: midodrine
Drug: Pyridostigmine Bromide — study 1 will be single blind. study 2 will be blinded randomized-control trial.
  Other Names: pyridostigmine
Drug: Mirabegron — study 1 will be single blind. study 2 will be blinded randomized-control trial.
Other: Placebo — placebo will only be used for study arm 2, the randomized blinded phase.
  Arms: Study 2

SUMMARY:
Dysregulation of blood pressure (BP), secondary to decentralized autonomic nervous system (ANS) control of the cardiovascular system, often results in chronic hypotension and orthostatic hypotension (OH) in persons with spinal cord injury (SCI), particularly in those with high cord lesions (i.e., above T6). While most hypotensive individuals with chronic SCI remain asymptomatic and do not complain of symptoms associated with cerebral hypoperfusion, evidence of reduced resting cerebral blood flow (CBF) has been reported in association with low systemic BP in the SCI and non-SCI populations. Reduced CBF in hypotensive individuals may lead to cognitive dysfunction, and we reported significantly impaired memory and marginally impaired attention processing in hypotensive individuals with SCI compared to a normotensive SCI cohort. Furthermore, we found that CBF was not increased during cognitive testing in individuals with SCI, which may contribute to impaired cognitive function compared to non-SCI controls. Although asymptomatic hypotension may have an adverse impact on cognitive function and quality of quality of life (QOL) clinical management of this condition is extremely low. In fact, we reported that while nearly 40% of Veterans with SCI were hypotensive, less than 1% carried the diagnosis of hypotension or were prescribed an anti-hypotensive medication. The discrepancy between incidence and treatment of asymptomatic hypotension in the SCI population may relate to a paucity of treatment options which are supported by rigorous clinical trials documenting safe and effective use of anti-hypotensive therapy on BP, CBF and cognitive function. We hypothesize these study medications may increase systolic blood pressure to the normal range and improve cerebral blood flow velocity. Results and conclusions will not be removed from the record.

DETAILED DESCRIPTION:
Study 1: Subjects will visit the laboratory between 3 and 9 times for 4 hours to determine the BP response to each dose of the 3 study medications (midodrine, pyridostigmine, and mirabegron). Upon arrival to the laboratory subjects will be randomized to receive midodrine, pyridostigmine, or mirabegron. Subjects will remain seated in their wheelchair for the duration of testing. Instrumentation will be applied by study personnel while subject is seated quietly, this can take up to 20 minutes. Instrumentation includes placement of 3 ECG electrodes for continuous HR monitoring and finger and brachial BP cuffs. BP, BR and HR will be recorded for 5-minutes before medication administration (baseline). After baseline, a small pill will be given with a glass of water. BP, BR and HR will be monitored for 5-minutes every 30 minutes for 4 hours after drug administration.

Study 2: Twenty will visit the laboratory on 4 occasions to determine the effects of three anti-hypotensive agents, compared to placebo, on BP, CBFv, and cognitive performance on selected neuropsychological tests. Upon arrival to the laboratory for every visit subjects will be randomized to receive midodrine, pyridostigmine, mirabegron, or matching placebo. Neither the study subject nor the investigator will know which is being administered. Subjects will remain seated in their wheelchair throughout the duration of the study session and will be closely monitored by study personnel. Instrumentation will include placement of 3 ECG electrodes for continuous heart rate (HR) monitoring, finger and brachial BP cuffs, and a Doppler ultrasound probe positioned at the left MCA for continuous CBFv monitoring. Subjects will remain quietly seated in their wheelchair for 30-minutes after instrumentation for a 5-minute recording of continuous HR, BP, and CBFv (baseline). Prior to the baseline data collection period, the first battery of cognitive tests will be administered. The study medication will be administered to the subject along with a glass of water approximately 30-minutes after arrival to the laboratory. There will be a 2 hour break period until the second cognitive battery begins.

ELIGIBILITY:
Inclusion Criteria:

Spinal Cord Injured

* Any level of injury
* Any ASIA grade of SCI
* Primarily wheelchair dependent for mobility
* Duration of injury ˃ 1 year

Exclusion Criteria:

* Current illness or infection
* History of severe autonomic dysreflexia (AD: condition where BP increases)
* More than 3 symptomatic events per week; BP elevations above 140/90 mmHg; adverse symptoms reporting (e.g., light headedness, dizziness, goosebumps, chills, nausea, etc.)
* Diagnosis of hypertension
* History of Traumatic Brain Injury (TBI)
* Documented history of traumatic brain injury (TBI)
* Neurological condition other than SCI (Alzheimer's disease, dementia, stroke, multiple sclerosis, Parkinson's disease, etc)
* History of epilepsy or other seizure disorder
* Liver or kidney disease
* Bladder problems including blockage of the urine and/or weak urine stream
* Diagnosis of a psychiatric disorder such as schizophrenia or bipolar disorder
* Diagnosis of artery disease, heart failure, irregular heartbeat, and AV block
* Allergies to aspirin, a yellow dye, pyridostigmine bromide, midodrine hydrochloride, lyethylene oxide, polyethylene glycol, hydroxypropyl cellulose, butylated hydroxytoluene, magnesium stearate, hypromellose, yellow ferric oxide, and red ferric oxide
* Had major surgery in the last 30 days
* Illicit drug abuse within the last 6 months
* Pregnant

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill M Wecht, Ed.D, Principal Investigator — James J. Peters VA Medical Center
Locations (2):
- United States (2):
  - Kessler Foundation Research Center, West Orange, New Jersey
  - James J Peters VAMC, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Study 1: Study 1 is a dose escalation, single blinded, trial to determine the individualized dose of each of 3 medications (midodrine, pyridostigmine, mirabegron) that increases systolic blood pressure (SBP) into the normal range (111-139 mmHg).
  Midodrine: 5 mg (Low), 10 mg (Medium), 15 mg (High) Mirabegron: 25 mg (Low), 50 mg (Medium), 75 mg (High) Pyridostigmine: 60 mg (Low), 90 mg (Medium), 120 mg (High) Within this dose escalation trial, each participant will be started on the lowest dose of each of the three medications, and may receive the medium or high dose depending on their SBP response.
  Study 2 is a randomized, placebo-controlled, double-blinded investigation to determine the effects of the normalization of SBP on cerebral blood flow, cognitive function, and quality of life. In study 2 participants will receive the dose of each medication that normalized their SBP in study 1.
  Midodrine: 5 mg (Low), 10 mg (Medium), 15 mg (High) Mirabegron: 25 mg (Low), 50 mg (Medium), 75 mg (High) Pyridostigmine: 60 mg (Low), 90 mg (Medium), 120 mg (High) Placebo In study 2 all participants will receive one dose (optimized for their SBP response) of each medication and placebo.
Period: Study 1
Arm/Group | Study 1
Started | 21
Midodrine (Low) | 19
Midodrine (Medium) | 6
Midodrine (High) | 0
Mirabegron (Low) | 19
Mirabegron (Medium) | 15
Mirabegron (High) | 8
Pyridostigmine (Low) | 19
Pyridostigmine (Medium) | 10
Pyridostigmine (High) | 5
Placebo | 0
Completed | 19
Not Completed | 2
Period: Study 2
Arm/Group | Study 1
Started | 18
Midodrine (Low) | 11
Midodrine (Medium) | 5
Midodrine (High) | 0
Mirabegron (Low) | 3
Mirabegron (Medium) | 7
Mirabegron (High) | 7
Pyridostigmine (Low) | 7
Pyridostigmine (Medium) | 5
Pyridostigmine (High) | 5
Placebo | 16
Completed | 16
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Study 1: Study 1 is a dose escalation, single blinded, trial to determine the individualized dose of each of 3 medications (midodrine, pyridostigmine, mirabegron) that increases systolic blood pressure (SBP) into the normal range (111-139 mmHg).
  Midodrine: 5 mg (Low), 10 mg (Medium), 15 mg (High) Mirabegron: 25 mg (Low), 50 mg (Medium), 75 mg (High) Pyridostigmine: 60 mg (Low), 90 mg (Medium), 120 mg (High) Within this dose escalation trial, each participant will be started on the lowest dose of each of the three medications, and may receive the medium or high dose depending on their SBP response.
  Study 2 is a randomized, placebo-controlled, double-blinded investigation to determine the effects of the normalization of SBP on cerebral blood flow, cognitive function, and quality of life. In study 2 participants will receive the dose of each medication that normalized their SBP in study 1.
  Midodrine: 5 mg (Low), 10 mg (Medium), 15 mg (High) Mirabegron: 25 mg (Low), 50 mg (Medium), 75 mg (High) Pyridostigmine: 60 mg (Low), 90 mg (Medium), 120 mg (High) Placebo In study 2 all participants will receive one dose (optimized for their SBP response) of each medication and placebo.
  Mirabegron: 25 mg (Low), 50 mg (Medium), 75 mg (High) Pyridostigmine: 60 mg (Low), 90 mg (Medium), 120 mg (High)
Arm/Group | Study 1
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.47 (10.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Description: Seated systolic blood pressure following intervention administration.
Time Frame: 4 hours
Population: Means are compared between medications and placebo of study 2, regardless of dose, as pre-specified in the study protocol.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Study 2: Placebo; Study 2: Midodrine; Study 2: Mirabegron; Study 2: Pyridostigmine: Study 2 is a blinded comparison of the seated systolic blood pressure responses to Midodrine Hydrochloride, Pyridostigmine Bromide, and Mirabegron compared to placebo in a randomized, double-blinded, placebo-control trial.
Arm/Group | Study 2: Placebo | Study 2: Midodrine | Study 2: Mirabegron | Study 2: Pyridostigmine
Number analyzed (Participants) | 16 | 16 | 16 | 16
mmHg | 93.21 (9.01) | 107.00 (11.07) | 95.8 (9.5) | 93.84 (9.69)

2. Primary Outcome: Number of Participants With Normal Blood Pressure Readings
Description: Number of participants with a systolic blood pressure readings between 111-139 mmHg in response to each of the four conditions:
  1. Placebo
  2. Midodrine
  3. Mirabegron
  4. Pyridostigmine
Time Frame: 4 hours
Population: Data are compared between medications and placebo of study 2, regardless of dose, as pre-specified in the study protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Study 2: Placebo: Study 2 is a blinded comparison of the seated systolic blood pressure responses to Midodrine Hydrochloride, Pyridostigmine Bromide, and Mirabegron compared to placebo in a randomized, double-blinded, placebo-control trial.
  Mirabegron: study 1 will be single blind. study 2 will be blinded randomized-control trial.
- Study 2: Midodrine: Study 2 is a blinded comparison of the seated systolic blood pressure responses to Midodrine Hydrochloride, Pyridostigmine Bromide, and Mirabegron compared to placebo in a randomized, double-blinded, placebo-control trial.
  Mirabegron: study 1 will be single blind. study 2 will be blinded randomized-control trial.
  Placebo: placebo will only be used for study arm 2, the randomized blinded phase.
- Study 2:Pyridostigmine: Study 2 is a blinded comparison of the seated systolic blood pressure responses to Midodrine Hydrochloride, Pyridostigmine Bromide, and Mirabegron compared to placebo in a randomized, double-blinded, placebo-control trial.
Arm/Group | Study 2: Placebo | Study 2: Midodrine | Study 2: Mirabegron | Study 2:Pyridostigmine
Number analyzed (Participants) | 16 | 16 | 16 | 16
Participants | 4 | 14 | 6 | 5

ADVERSE EVENTS:
Time Frame: For the duration of the study (4-hours).
Description: Risks of AE, SAE, and all cause mortality were assessed for each medication/dose regardless of the study arm, as per the protocol.
Groups:
- Midodrine (Low); Midodrine (Mid); Midodrine (High); Mirabegron (Low); Mirabegron (Mid); Mirabegron (hi); Pyridostigmine (Low); Pyridostigmine (Mid); Pyridostigmine (hi): Study 1 and 2
- Placebo: Study 2
Arm/Group | Midodrine (Low) | Midodrine (Mid) | Midodrine (High) | Mirabegron (Low) | Mirabegron (Mid) | Mirabegron (hi) | Pyridostigmine (Low) | Pyridostigmine (Mid) | Pyridostigmine (hi) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/6 | 0/0 | 0/19 | 0/15 | 0/8 | 0/19 | 0/10 | 0/5 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/6 | 0/0 | 0/19 | 0/15 | 0/8 | 0/19 | 0/10 | 0/5 | 0/16
Other Adverse Events (participants affected / at risk) | 0/19 | 0/6 | 0/0 | 0/19 | 0/15 | 0/8 | 0/19 | 0/10 | 0/5 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT02893553/Prot_SAP_ICF_000.pdf